CLINICAL TRIAL: NCT04599725
Title: TelAbortion: Medical Abortion by Direct-to-patient Telemedicine and Mail
Brief Title: Feasibility of Telemedicine Medical Abortion
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Other Study IDs: 1049
Record Dates: First submitted 2020-10-19; First posted 2020-10-23 (Actual); Last update posted 2022-02-04 (Actual); Status verified 2020-10

CONDITIONS: Pregnancy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Pregnant people
  Interventions: Drug: medical abortion

INTERVENTIONS:
Drug: medical abortion — medical abortion

SUMMARY:
This pilot study is designed to obtain data on the safety, acceptability, and feasibility of providing abortion by direct-to-patient telemedicine and mail.

ELIGIBILITY:
Inclusion Criteria:

* desires abortion

Exclusion Criteria:

* medically ineligible for procedure

Ages: 10 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: People seeking abortion
Sampling Method: Non-Probability Sample
Enrollment: 413 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raymond, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (15):
- United States (15):
  - Planned Parenthood of the Rocky Mountains, Denver, Colorado
  - Carafem, Washington D.C., District of Columbia
  - Carafem, Atlanta, Georgia
  - The University of Hawaii Women's Options Centers, Honolulu, Hawaii
  - Carafem, Skokie, Illinois
  - Emma Goldman Clinic, Iowa City, Iowa
  - Maine Family Planning, Augusta, Maine
  - Carafem, Chevy Chase, Maryland
  - Maine Family Planning, Boston, Massachusetts
  - Planned Parenthood Minnesota, North Dakota, South Dakota, Saint Paul, Minnesota
  - Planned Parenthood of Montana, Billings, Montana
  - Planned Parenthood of the Rocky Mountains, Albuquerque, New Mexico
  - Maine Family Planning, New York, New York
  - Planned Parenthood Columbia Willamette, Portland, Oregon
  - Planned Parenthood Columbia Willamette, Vancouver, Washington